CLINICAL TRIAL: NCT05783232
Title: Radicle™ Health1: A Randomized, Blinded, Placebo-controlled Study of Health and Wellness Formulations and Their Effects on Overall Health
Brief Title: Radicle Health1: A Study of Health and Wellness Formulations and Their Effects on Overall Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-22D07
Record Dates: First submitted 2023-03-08; First posted 2023-03-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Sleep; Pain; Depression; Anxiety
MeSH Terms: conditions — Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arm
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Control 1 Capsules (Placebo Comparator): Health Product Form 1 Capsules - control
  Interventions: Dietary Supplement: Placebo Control Form 1 Capsules
- Active Product 1.1 Capsules (Experimental): Health Product Form 1 Capsules - active product 1
  Interventions: Dietary Supplement: Health Active Study Product 1.1 Capsules
- Active Product 1.2 Capsules (Experimental): Health Product Form 1 Capsules - active product 2
  Interventions: Dietary Supplement: Health Active Study Product 1.2 Capsules
- Active Product 1.3 Capsules (Experimental): Health Product Form 1 Capsules - active product 3
  Interventions: Dietary Supplement: Health Active Study Product 1.3 Capsules

INTERVENTIONS:
Dietary Supplement: Placebo Control Form 1 Capsules — Participants will use their Placebo Control Form 1 Capsules as directed for a period of 4 weeks.
  Arms: Placebo Control 1 Capsules
Dietary Supplement: Health Active Study Product 1.1 Capsules — Participants will use their Radicle Health Active Study Product 1.1 Capsules as directed for a period of 4 weeks.
  Arms: Active Product 1.1 Capsules
Dietary Supplement: Health Active Study Product 1.2 Capsules — Participants will use their Radicle Health Active Study Product 1.2 Capsules as directed for a period of 4 weeks.
  Arms: Active Product 1.2 Capsules
Dietary Supplement: Health Active Study Product 1.3 Capsules — Participants will use their Radicle Health Active Study Product 1.3 Capsules as directed for a period of 4 weeks.
  Arms: Active Product 1.3 Capsules

SUMMARY:
A randomized, blinded, placebo-controlled study of health and wellness product formulations and their effects on overall health

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with adult participants, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for better health during screening; (2) indicate an interest in taking a health and wellness product to potentially help improve their health, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data will be collected electronically from eligible participants over 5 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Resides in the United States
* Endorses: a desire for better sleep and/or focus, less pain, less feelings of stress, depression, and/or anxiety, and/or more energy (less fatigue)
* Expresses a willingness to take a study product that may contain cannabinoids (or placebo) and not know the product identity until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid physical shipping address and mobile phone number
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Reports current enrollment in a clinical trial
* The QOL score greater than 5 during enrollment
* Unable to read and understand English
* Lack of reliable daily access to the internet
* Reports taking any medication that warns against grapefruit consumption
* Reports current or recent (within 3 months) use of chemotherapy, immunotherapy, or oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1494 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Change in overall health-related quality of life | 4 weeks
  Mean difference in overall health score as assessed by Patient Reported Outcome Measurement System (PROMIS) 29+2 Profile (PROPr; scale 70-120; with higher scores corresponding to greater overall health across 7 health domains: physical function, ability to participate in social roles and activities, cognitive function, anxiety, depression, fatigue, sleep disturbance, pain interference and pain intensity)

SECONDARY OUTCOMES:
Change in physical function | 4 weeks
  Mean difference in physical function score as assessed by PROMIS PROPr items related to physical function (scale 4-20; with higher scores corresponding to greater physical function)
Change in feelings of anxiety | 4 weeks
  Mean difference in feelings of anxiety score as assessed by PROMIS PROPr items related to anxiety (scale 4-20; with higher scores corresponding to more severe feelings of anxiety)
Change in feelings of depression | 4 weeks
  Mean difference in feelings of depression score as assessed by PROMIS PROPr items related to depression (scale 4-20; with higher scores corresponding to more severe feelings of depression)
Change in fatigue | 4 weeks
  Mean difference in fatigue score as assessed by PROMIS PROPr questions related to fatigue (scale 4-20; with higher scores corresponding to more severe fatigue)
Change in sleep disturbance | 4 weeks
  Mean difference in sleep disturbance score as assessed by PROMIS PROPr items related to sleep disturbance (scale 4-20; with higher scores corresponding to greater sleep disturbance)
Change in socialization ability | 4 weeks
  Mean difference in socialization ability score as assessed by PROMIS PROPr items related to (scale 4-20; with higher scores corresponding to greater ability to participate in social roles and activities)
Change in pain | 4 weeks
  Mean difference in pain score as assessed by PROMIS PROPr items related to pain (scale 1-15; with higher scores corresponding to greater pain)
Change in cognitive function | 4 weeks
  Mean difference in cognitive function score as assessed by PROMIS PROPr items related to cognitive function (scale 2-10; with higher scores corresponding to greater cognitive function)
Change in libido | 4 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 2-10; where higher scores correspond to greater interest in sexual activities)
Minimal clinical importance difference (MCID) in overall health-related quality of life | 4 weeks
  Likelihood of achieving a MCID in overall health-related quality of life, as measured by PROMIS PROPr (scale 70-120; with higher scores corresponding to greater overall health-related quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com